CLINICAL TRIAL: NCT00517270
Title: High-dose Proton Pump Inhibitor for the Treatment of Gastro-oesophageal Reflux Related Non-cardiac Chest Pain - a Randomized Double-blind Placebo-controlled Study.
Brief Title: A Study of the Use of High-dose Proton Pump Inhibitor for the Treatment of Gastro-oesophageal Reflux Related Non-cardiac Chest Pain - a Randomized Double-blind Placebo-controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC1932-02; HARECCTR0500032
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Chest Pain
Keywords: Non-cardiac chest pain
MeSH Terms: conditions — Chest Pain | interventions — Rabeprazole

INTERVENTIONS:
Drug: Rabeprazole 20mg twice daily

SUMMARY:
Non-cardiac chest pain accounts for 2-5% of all emergency presentations. In the United States, it has been estimated approximately that US$8 billion was spent annually for the initial care of patients suspected to have an acute coronary syndrome, but who were subsequently found not to have coronary artery disease (1). The most common cause of non-cardiac chest pain is gastro-oesophageal reflux disease (2). Two randomized, double-blind, placebo-controlled trials on the use of omeprazole versus placebo for the treatment of NCCP have been published in the western population and reported an efficacy of 62% to 80% (3,4). High-dose omeprazole was used in the previous trials (3,4). Recently, it has been shown that rabeprazole, which is a newly developed benzimidazole proton pump inhibitor, is a more potent and rapid inhibitor of H+,K+-ATPase and acid secretion than omeprazole, lansoprazole and pantoprazole (5,6). Whether the above findings applied to Chinese population is unknown. Thus we would like to propose a randomized double-blind placebo-controlled trial to study the effects of high-dose proton pump inhibitor for the treatment of non-cardiac chest pain in Chinese population. The aim of this study is to evaluate the efficacy of high-dose proton pump inhibitor for the treatment of gastro-oesophageal reflux related non-cardiac chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients with age over 18 years old
* Patients with chest pain for at least 12 weeks, in the preceding 12 months who are evaluated by cardiac catheterization or exercise radionuclide scan / persantin radionuclide scan will be assessed for suitability to enter the study. Patients will be included if the results of the cardiac investigation are normal.

Exclusion Criteria:

* Patients with history of significant cardiac, renal, pulmonary or hepatic diseases.
* Patients with history of gastrointestinal surgery or peptic ulcer diseases.
* Intake of H2 receptor blockers, bismuth or proton pump inhibitors or drugs affecting gastrointestinal motility in the preceding four weeks.
* Patients who are pregnant or lactating.
* Patients who are suffering from costochrondritis.
* Patients who are known to be sensitive to proton pump inhibitor.
* Patients with glaucoma and benign prostatic hypertrophy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2003-03; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
Symptoms assessment, quality of life. | 12 Weeks

SECONDARY OUTCOMES:
Compliance | 4 Weeks
Adverse effects | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ting Kin Cheung, Dr, Principal Investigator — Department of Medicine, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China